CLINICAL TRIAL: NCT05672615
Title: Mood Alterations in the Patients With Non-Muscle Invasive Bladder Cancer Treated With Bacillus Calmete-Guerin
Brief Title: Mood Alterations in the Patients With Non-Muscle Invasive Bladder Cancer Treated With BCG
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00306420
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Bacillus Calmette-Guerin; Mood Alterations
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Surveys and Questionnaires; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked for research blood and urine samples prior to the start of treatment and throughout the treatment course. The study team will also ask participants permission to utilize excess tissue from standard of care procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Muscle Invasive Bladder Cancer - Bacillus Calmete-Guerin (BCG) intravesical treatments: Participants who are receiving BCG intravesical treatments will be asked to provide research urine samples and blood samples prior to and during their treatment course. Participants will also be asked to complete the Zung Self-Rating Anxiety Scale and Zung Self-Rating Depression Scale at the start and throughout the treatment course. Participants will be given a daily mood diary to complete at the following timepoints: 6-week induction treatment, 3-week maintenance treatment, and the 3-month follow-up. The study team will ask permission from participants to utilize excess tissue samples from standard of care procedures and biopsies. Participants' medical history and clinical data will also be collected for the study.
  Interventions: Other: Questionnaires; Other: Daily Mood Diaries; Other: Urine Specimen Collection; Other: Research Blood Draw; Other: Utilize excess tissue from a standard of care procedure
- Non-Muscle Invasive Bladder Cancer - Chemotherapy intravesical treatments: Participants who are receiving chemotherapy intravesical treatments will be asked to provide research urine samples and blood samples prior to and during their treatment course. Participants will also be asked to complete the Zung Self-Rating Anxiety Scale and Zung Self-Rating Depression Scale at the start and throughout the treatment course. Participants will be given a daily mood diary to complete at the following timepoints: 6-week induction treatment, 3-week maintenance treatment, and the 3-month follow-up. The study team will ask permission from participants to utilize excess tissue samples from standard of care procedures and biopsies. Participants' medical history and clinical data will also be collected for the study.
  Interventions: Other: Questionnaires; Other: Daily Mood Diaries; Other: Urine Specimen Collection; Other: Research Blood Draw; Other: Utilize excess tissue from a standard of care procedure

INTERVENTIONS:
Other: Questionnaires — Participants will be given the Zung Self-Rating Anxiety Scale and Zung Self-Rating Depression Scale to complete prior to each induction intravesical treatment and prior to 3-month follow-up appointments.
Other: Daily Mood Diaries — Participants will be given daily mood diaries to complete during their 6-week induction intravesical treatment, 3-week maintenance treatment course, and between 3-month follow-up appointments.
Other: Urine Specimen Collection — Urine collections from patients will occur prior to each induction intravesical treatment and at 3-month follow-up cystoscopy appointments. An at home urine collection may occur 6 hours post intravesical treatment.
Other: Research Blood Draw — Blood collections will occur prior to first intravesical treatment, prior to fourth intravesical treatment, and each 3-month cystoscopy as indicated by the participant's treatment course.
Other: Utilize excess tissue from a standard of care procedure — Participants may indicate permission to provide excess tissue from a clinically indicated procedure for research purposes.

SUMMARY:
The purpose of this study is to evaluate mood changes in patients with Non-Muscle Invasive Bladder Cancer who are receiving intravesical Bacillus Calmete-Guerin (BCG). Patients with Non-Muscle Invasive Bladder Cancer receiving intravesical treatments are eligible to participate in this study. Participation involves providing research blood and urine samples prior to the start of treatment and throughout the treatment course. The study team will also collect participant's medical history and clinical information. Participants will be asked to complete questionnaires and daily mood diaries.

DETAILED DESCRIPTION:
Patients with Non-Muscle Invasive Bladder Cancer who are receiving intravesical treatments are eligible to participate in this study. Participants will be asked to complete the Zung Self-Rating Anxiety Scale and Zung Self-Rating Depression Scale prior to each induction intravesical treatment. During the 6-week induction intravesical treatment, participants will also be given a daily mood dairy to complete. Urine Specimens will be collected prior to each induction intravesical treatment and at each 3-month cystoscopy appointment during the treatment course. An at home urine collection may occur 6 hours post intravesical treatment. Research Blood Samples will be collected prior to the first induction intravesical treatment, prior to the fourth intravesical treatment, and prior to each 3-month follow-up cystoscopy as indicated by the participant's treatment course. Participants will be asked to complete the Zung Self-Rating Anxiety Scale and Zung Self-Rating Depression Scale prior to each 3-month follow-up cystoscopy during the treatment course. A 3-week daily mood diary will be completed by participants during the 3-week intravesical maintenance treatment. Participants will be given a daily mood diary to complete between the 3-month follow-up cystoscopy appointments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a pathologically confirmed non-muscle invasive bladder cancer
* Age ≥ 18 years old
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients that are not candidates for intravesical treatment due to the nature of their disease, such as variant histology or progressive disease after a prior course of intravesical treatment.
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that are 18 years old or older who have pathologically confirmed non-muscle invasive bladder cancer. Subjects receiving intravesical treatments as part of their standard of care.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in cytokine response as assessed by urine samples | Prior to each 6-week intravesical treatment and every 3-month Cystoscopy for 24 months
  Collect urine samples from the patients with non-muscle invasive bladder cancer who are undergoing intravesical instillations for cytokine response to treatment
Change in cytokine response as assessed by blood samples | Prior to the first intravesical treatment, prior to the fourth intravesical treatment, and prior to the each 3-month follow-up cystoscopy
  Collect blood samples from the patients with non-muscle invasive bladder cancer who are undergoing intravesical instillations for cytokine response to treatment
Screening for Mood Disorders utilizing the Zung Self Rating Depression Scale | Prior to each induction intravesical treatment for six weeks and each 3-month surveillance visit
  Screen for mood disorders in patients diagnosed with Non-muscle Invasive Bladder Cancer at baseline and while undergoing treatment utilizing the Zung Self Rating Depression Scale. The Zung Self-Rating Depression Scale has the following score ranges: Normal Range (25-49), Mildly Depressed (50-59), Moderately Depressed (60-69), Severely Depressed (70 and above)

SECONDARY OUTCOMES:
Screening for Mood Disorders utilizing the Zung Self Rating Anxiety Scale | Prior to each induction intravesical treatment for six weeks and each 3-month surveillance visit
  Screen for mood disorders in patients diagnosed with Non-muscle Invasive Bladder Cancer at baseline and while undergoing treatment utilizing the Zung Self Rating Anxiety Scale
Screening for Mood Disorders utilizing daily mood diaries | Daily mood diary for 6-week induction intravesical treatment course, daily mood diary for 3-week intravesical treatment maintenance course, and daily mood diary between 3-month follow up cystoscopy appointments
  Screening for Mood Disorders at baseline and through the treatment course with daily mood diaries
Evaluate DNA and RNA-based liquid biopsy biomarkers and correlate them with tissue response | Prior to the first intravesical treatment, prior to the fourth intravesical treatment, and prior to each 3-month follow-up cystoscopy
  Collect blood and urine samples from the patients with non-muscle invasive bladder cancer who are undergoing intravesical instillations and compare them with excess tissue from a clinically indicated procedure

CONTACTS AND LOCATIONS:
Overall Officials: Armine Smith, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sibley Memorial Hospital, Washington D.C., District of Columbia, United States